CLINICAL TRIAL: NCT06541197
Title: The Effect of Adding Functional Electrical Stimulation Bicycle Ergometry to Robotic Rehabilitation on Walking Function and Lower Extremity Functional Recovery in Patients With Chronic Incomplete Spinal Cord Injury
Brief Title: The Effect of Functional Electrical Stimulation Cycling Ergometry in Addition to Robotic Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Örücü Atar, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AESH-EK1-2024-0088
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; functional electrical stimulation bicycle ergometry; robotic rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic rehabilitation combined with Functional Electrical Stimulation (FES) bicycle ergometry group (Active Comparator): Robotic assisted walking exercise will be performed in the walking exercise robot for a total of 20 sessions for 4 weeks. For FES bicycle ergometry, a current-controlled six-channel stimulator (RT 300-SLSA; Restorative Therapies, Baltimore, MD, USA) will be used. The quadriceps, hamstring and tibialis anterior muscles will be stimulated bilaterally with six channels through 3 × 4 cm2 adhesive surface electrodes. Stimulation intensity will be adjusted according to palpable muscle contraction and sensory discomfort felt by patients with incomplete SCI. The pedaling cadence range will be set to 40-50 rotations per minute. Robotic rehabilitation will be applied in 30-minute sessions with Lokomat v5 (Hocoma, Volketswil, Switzerland) device for lower extremity rehabilitation. FES bicycle ergometry will be performed in 30-minute sessions for 4 weeks for a total of 20 sessions under the supervision of a physician before robotic rehabilitation.
  Interventions: Other: Robotic rehabilitation combined with Functional Electrical Stimulation (FES) bicycle ergometry group
- Robotic rehabilitation (Active Comparator): Robotic rehabilitation will be applied in 30-minute sessions with Lokomat v5 (Hocoma, Volketswil, Switzerland) device for lower extremity rehabilitation. Robotic assisted walking exercise will be performed in the walking exercise robot for a total of 20 sessions for 4 weeks.
  Interventions: Other: Robotic rehabilitation

INTERVENTIONS:
Other: Robotic rehabilitation combined with Functional Electrical Stimulation (FES) bicycle ergometry group — Robotic rehabilitation will be applied in 30-minute sessions with Lokomat v5 (Hocoma, Volketswil, Switzerland) device for lower extremity rehabilitation. Robotic assisted walking exercise will be performed in the walking exercise robot for a total of 20 sessions for 4 weeks. For FES bicycle ergometry, a current-controlled six-channel stimulator (RT 300-SLSA; Restorative Therapies, Baltimore, MD, USA) will be used. The quadriceps, hamstring and tibialis anterior muscles will be stimulated bilaterally with six channels through 3 × 4 cm2 adhesive surface electrodes. Stimulation intensity will be adjusted according to palpable muscle contraction and sensory discomfort felt by patients with incomplete SCI. The pedaling cadence range will be set to 40-50 rotations per minute. FES bicycle ergometry will be performed in 30-minute sessions for 4 weeks for a total of 20 sessions before robotic rehabilitation.
  Arms: Robotic rehabilitation combined with Functional Electrical Stimulation (FES) bicycle ergometry group
Other: Robotic rehabilitation — Robotic rehabilitation will be applied in 30-minute sessions with Lokomat v5 (Hocoma, Volketswil, Switzerland) device for lower extremity rehabilitation. Robotic assisted walking exercise will be performed in the walking exercise robot for a total of 20 sessions for 4 weeks.
  Arms: Robotic rehabilitation

SUMMARY:
Spinal cord injury (SCI) is a devastating neurological condition resulting from either traumatic or non-traumatic causes, leading to loss of motor, sensory, and autonomic functions in individuals. Statistics indicate that more than 75% of individuals with incomplete SCI regain some degree of ambulatory function.

Authors' aim in this study is to investigate the effect of adding functional electrical stimulation (FES) bicycle ergometry to robotic rehabilitation on lower extremity functional recovery and ambulation in patients with chronic incomplete SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a devastating neurological condition resulting from either traumatic or non-traumatic causes, leading to loss of motor, sensory, and autonomic functions in individuals. Statistics indicate that more than 75% of individuals with incomplete SCI regain some degree of ambulatory function. To the authors' knowledge, no other study has investigated the effect of adding FES bicycle ergometry to robotic rehabilitation on lower extremity functional recovery and ambulation in patients with chronic incomplete SCI. Authors' hypothesis is that the group receiving FES bicycle ergometry in addition to robotic rehabilitation will achieve better functional recovery and ambulation compared to the group receiving only robotic rehabilitation. In this context, authors' aim in this study is to investigate the effect of adding functional electrical stimulation bicycle ergometry to robotic rehabilitation on lower extremity functional recovery and ambulation in patients with chronic incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Motor Incomplete spinal cord injury (ASIA C and D).
2. At least 6 months post spinal cord injury.
3. Age between 18 and 65 years.
4. Ability to walk at least 10 meters independently or with assistive devices such as a cane or crutches.
5. Signed informed consent form indicating willingness to participate in the study.

Exclusion Criteria:

1. Severe spasticity or joint contracture in the lower extremities that impedes movement.
2. Presence of metallic implants in the lower extremities.
3. Stage 2 or higher pressure ulcers on the sacral or coccygeal regions.
4. Co-existing peripheral neuropathy.
5. Permanent urinary catheter use.
6. Contraindications for walking exercises (e.g., cognitive impairment preventing exercise compliance, unstable epilepsy or unexplained convulsions, unstable acute cardiac arrhythmia or heart failure, presence of a cardiac pacemaker).
7. Psychiatric disorders or cognitive problems that prevent completing questionnaires and assessment scales.
8. Presence of other neurological or muscular diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Walking Index for Spinal Cord Injury (WISCI II) | at baseline and change from baseline WISCI II at 4 weeks
  An index that evaluates walking ability post-SCI, scoring from 0 to 20 based on the need for personal assistance, use of orthoses, walkers, crutches, canes, or no assistive devices. Scores for the WISCI II scale range from 0 to 20 (0: most severe impairment, 20: mild impairment).

SECONDARY OUTCOMES:
Lower Extremity Motor Score (LEMS) | at baseline and change from baseline LEMS at 4 weeks
  A method for determining muscle strength in key motor muscles of the lower extremities according to the ASIA impairment scale. (0) No observable or palpable muscle contraction. (1) Observable or palpable muscle contraction, but no joint movement. (2) Completes joint movement when gravity is eliminated. (3) Completes joint movement against gravity, but no resistance. (4) Completes joint movement against moderate resistance. (5) Completes joint movement against full resistance. Total score for the LEMS scale range from 0 to 50.
Spinal Cord Independence Measure (SCIM) | at baseline and change from baseline SCIM at 4 weeks
  An assessment tool for physical disabilities and independence in daily living activities for SCI patients. It consists of three main sections: self-care, respiration and sphincter control, and mobility, with a total score ranging from 0 to 100 (higher scores indicate greater independence).
Ten (10)-Meter Walk Test | at baseline and change from baseline 10-meter walk test at 4 weeks
  A measure of ambulation where the patient walks a 10-meter distance at a normal pace, and the time taken is recorded.
Two (2)-Minute Walk Test | at baseline and change from baseline 2-minute walking test at 4 weeks
  Measure of functional capacity where the patient walks the maximum distance possible in 2 minutes on a marked 30-meter flat and firm surface. The 2-minute walk test is a safe alternative to the 6-minute walk test, particularly in SCI patients, as it shows a strong correlation with it.
Timed Up and Go Test (TUGT) | at baseline and change from baseline TUGT at 4 weeks
  An evaluation of mobility where patients are asked to rise from a chair, walk a 3-meter distance, return, and sit down, with the time taken recorded. Assistive devices may be used if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Örücü Atar, MD, Principal Investigator — Associate professor
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No